CLINICAL TRIAL: NCT04870112
Title: A Phase 1/2a, Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of Subcutaneous Durvalumab in Patients With Non-Small Cell and Small Cell Lung Cancer - SCope-D1
Brief Title: A Study to Evaluate Subcutaneous Durvalumab in Patients With Non-Small Cell Lung Cancer and Small Cell Lung Cancer
Acronym: SCope-D1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: AstraZeneca has decided to stop further enrollment and the study was terminated when all patients in Part 1 completed their last study visit. No safety issues or clinical concerns however, have been identified for this study. Part 2 was not initiated
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9072C00001; 2020-006041-18 (EudraCT Number)
Record Dates: First submitted 2021-04-16; First posted 2021-05-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: imfinzi; durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — durvalumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with NSCLC (Experimental): Patients with Non-Small Cell Lung Cancer
  Interventions: Drug: Durvalumab
- Patients with SCLC (Experimental): Patients with Small Cell Lung Cancer
  Interventions: Drug: Durvalumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Durvalumab — Anti-PD-L1 antibody
  Other Names: MEDI4736, IMFINZI
Drug: Cisplatin — Chemotherapy
  Arms: Patients with SCLC
Drug: Carboplatin — Chemotherapy
  Arms: Patients with SCLC
Drug: Etoposide — Chemotherapy
  Arms: Patients with SCLC

SUMMARY:
This study has 2 parts: dose finding and dose confirmatory.

In Part 1, the dose finding phase of the study, there will be 3 or more dosing levels to find out what dose of durvalumab administered as an infusion under the skin acts similarly to durvalumab administered into a vein. 24 participants with Non-Small Cell Lung Cancer will be enrolled for a 12 month treatment period and 3 months follow up

In Part 2, the dose confirmation phase of the study, participants will receive the dose of durvalumab identified in Part 1 of the study. The goal of Part 2 will be to learn more about the way that the body processes durvalumab when administered as an infusion under the skin. Approximately 90 participants with Non-Small Cell Lung Cancer will be enrolled; additionally, up to 10 participants with Small Cell Lung Cancer (who will receive concurrent chemotherapy) will be enrolled for a 12 treatment period and a 3 month follow-up period.

AstraZeneca has decided to stop further enrollment and the study was terminated when all patients in Part 1 (Phase I) completed their last study visit. No safety issues or clinical concerns however, have been identified for this study. Part 2 (Phase II) was not initiated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented unresectable Stage III NSCLC that has not progressed following definitive platinum based CRT or extensive disease (Stage IV) SCLC
* ECOG performance status of 0 or 1
* For participants with SCLC: At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 TL at baseline
* Absence of EGFR mutation or ALK rearrangement prior to screening

Exclusion Criteria:

* History of allogeneic organ transplantation
* Autoimmune or inflammatory disorders, diverticulitis, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome
* Uncontrolled intercurrent illness
* History of another primary malignancy
* History of active primary immunodeficiency
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Brain metastases or spinal cord compression
* Persistent toxicities (CTCAE Grade >2) caused by previous anticancer therapy, excluding alopecia
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Observed serum concentration (Ctrough) | Approximately 16 months
Number of patients with injection site reactions and immune-mediated reactions | Approximately 16 months
Maximum observed serum concentration (Cmax) | Approximately 16 months

SECONDARY OUTCOMES:
Time to maximum observed serum concentration (tmax) of durvalumab | Approximately 16 months
Area under the Plasma Concentration versus Time Curve (AUCτ) of durvalumab | Approximately 16 months
Incidence of Adverse Events | Approximately 16 months
Changes in WHO/ECOG performance status | Approximately 16 months
Occurrence of abnormal ECG - PR, QRS, QT, and QT interval corrected by Fridericia's formula intervals | Approximately 16 months
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by abnormality in clinical chemistry | Approximately 16 months
  Clinical chemistry will be assessed by liver function(Alanine aminotransferase, Aspartate aminotransferase, albumin, total bilirubin), kidney function (e.g. Urea, Creatinine) and endocrine function(TSH, T3 free,T4 free)
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by abnormality in haematology | Approximately 16 months
  Hematology will be assessed by white cell count, platelet count, absolute neutrophil count and absolute lymphocyte count.
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by vital signs (blood pressure in mmHg) | Approximately 16 months
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by vital signs (pulse rate) in beats per minute | Approximately 16 months
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by vital signs (respiration rate) in breaths per minute | Approximately 16 months
Safety and tolerability of SC dosing of durvalumab in participants with unresectable stage III NSCLC as assessed by vital signs (temperature) in degrees Celsius | Approximately 16 months
Incidence of of anti-drug antibodies (ADA) and neutralizing antibodies | Approximately 16 months
Part 2 only: Overall Response Rate (ORR) - proportion of participants with a complete or partial response to treatment as determined using RECIST 1.1 guidelines | Approximately 16 months
Part 2 only: Best Objective Response (BoR) - participant's best response following first dose of study drug | Approximately 16 months

OTHER OUTCOMES:
Incidence of injection site reactions reported through ISQ Symptoms questionnaire | Approximately 16 months
Treatment satisfaction reported using ISQ Satisfaction questionnaire | Approximately 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Suli Bolus, MD, Study Director — AstraZeneca
Locations (7):
- United States (2):
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Christchurch, New Zealand
- Spain (2):
  - Research Site, Badalona
  - Research Site, Majadahonda
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: AstraZenecaClinicaltrials.com — https://www.astrazenecaclinicaltrials.com/study/D9072C00001/